CLINICAL TRIAL: NCT03163147
Title: The Effect and Frequency of Helicobacter Pylori Infection in Primary Immune Thrombocytopenic Patients Not Respond on Steroid Therapy.
Brief Title: The Effect and Frequency of Helicobacter Pylori Infection in Primary Immune Thrombocytopenic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Badr, Assiut University, Assiut University
Other Study IDs: assiut 5000
Record Dates: First submitted 2017-05-14; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Effects Toxics
Keywords: frequency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immune thrombocytopenia (ITP) is an autoimmune disorder characterized by low platelet count (i.e less than 100.000) . In ITP, platelet surface membrane proteins become antigenic for unknown reasons , leading to stimulation of the immune system , autoantibody production, and platelet destruction In recent years ,the list of etiologies of ITP has been steadily increasing, so the term "idiopathic" is becoming obsolete, increasingly replaced by "immune"TP .

Treatment of ITP may be conceptually divided into rescue therapy and maintenance therapy . the terminology of corticosteroid-dependence means The need for ongoing or repeated doses administration of corticosteroids for at least 2 months to maintain a platelet count at or above 30 _ 109/L and/or to avoid bleeding. So, patients with corticosteroid dependence are considered non responders

DETAILED DESCRIPTION:
• Immune thrombocytopenia (ITP) is an autoimmune disorder characterized by low platelet count (i.e less than 100.000) . In ITP, platelet surface membrane proteins become antigenic for unknown reasons , leading to stimulation of the immune system , autoantibody production, and platelet destruction In recent years ,the list of etiologies of ITP has been steadily increasing, so the term "idiopathic" is becoming obsolete, increasingly replaced by "immune"TP.

Treatment of ITP may be conceptually divided into rescue therapy and maintenance therapy. the terminology of corticosteroid-dependence means The need for ongoing or repeated doses administration of corticosteroids for at least 2 months to maintain a platelet count at or above 30 _ 109/L and/or to avoid bleeding. So, patients with corticosteroid dependence are considered non responders The recent entry of Helicobacter pylori to the growing list of etiologies of itp has stirred much interest. . The relationship between H pylori infection and immune thrombocytopenia (ITP) is less clear .

However, among patients with H.pylori-associated ITP, a significant percentage achieve lasting remission after eradication of H.pylori .

H.pylori can be readily detected by non invasive methods, the C-urea breath test and antigen detection in stools are considered to be the most accurate, with both sensitivity and specificity in the range of 90% to 95% .

ELIGIBILITY:
Inclusion Criteria:

1.Patients diagnosed ITP and failed on steroid therapy.

Exclusion Criteria:

1. Patients with systemic lupus erythromatous
2. Drug administration
3. Hepatitis c infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: . Detect the frequency of H pylori infection in patients diagnosed itp not respond on steroid therapy 2. Detect the effect of H pylori in those patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of primary thrombocytopenic patients with helicobacter pylori infection who recieved its treatment and improved clinically and laboratory. | one year

IPD SHARING:
Plan to Share IPD: No